CLINICAL TRIAL: NCT06399341
Title: PAPILOBS GR: A Clinical Investigation to Assess the Effectiveness of PAPILOCARE® in the Regression of Cervix Cytological Abnormalities Caused by HPV.
Brief Title: Clinical Effectiveness of PAPILOCARE® in Regression of Cervix HPV Cytological Abnormalities (PAPILOBS GR).
Acronym: PAPILOBSGR
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-PPL-EL-130
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult women with ASCUS or LSIL result in routine Pap-test.: Adult HPV-positive women with Atypical Squamous Cells of Undetermined Significance (ASCUS) or Low-grade Squamous Intraepithelial Lesions (LSIL) cervical cytology with concordant colposcopy were treated with Papilocare for 6 months (1 cannula/day for 21 days during first month + 1 cannula/alternate days for subsequent 5 months), extending to a total of 12 months if needed.
  Interventions: Device: Papilocare vaginal gel

INTERVENTIONS:
Device: Papilocare vaginal gel — Treatment with Papilocare® for 6 months (1 cannula/day for 21 days during first month + 1 cannula/alternate days for subsequent 5 months)

SUMMARY:
The present study is a multicenter, open, non-interventional, prospective observational clinical study for the evaluation of the effectiveness of Papilocare® (medical device with CE mark) in the regression of cervix cytological abnormalities caused by HPV.

DETAILED DESCRIPTION:
524 participants were enrolled in the study from approximately 44 Greek sites. At baseline (Visit 1) written informed consent was obtained, participants' eligibility criteria were checked and medical history data were collected. Participants were advised to be treated with Papilocare® for 6 months (1 cannula/day for 21 days during first month + 1 cannula/alternate days for subsequent 5 months). At 6 months (Visit 2) primary and secondary objectives were evaluated. If needed and based on physician's decision, treatment was extended to a total of 12 months (Visit 3) and primary and secondary endpoints were evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

Women over 18 years of age who have been or not vaccinated against HPV.

1. Able to read and understand the Informed Consent Form and agree to participate in the study by signing the Informed Consent Form.
2. Patients with ASCUS or LSIL routine cytological examination and positive High Risk (HR) HPV molecular test, up to 3 months before inclusion in the study.
3. Patients who, due to this condition, undergo a colposcopy and have a concordant result with cytology.

Exclusion Criteria:

1. Any gynecological or non-gynecological condition / lesion / pathology for which, according to clinical judgment, the use of Papilocare® is not recommended or its use has contraindications.
2. Fertile women who do not use effective contraceptive methods, pregnant women, women with suspected pregnancy or intention to become pregnant within the next 6 months, or breastfeeding women.
3. Women who use vaginal contraceptives or other vaginal hormone treatments during the study.
4. Participation in another clinical trial either currently or 4 weeks before enrolling in the study.
5. Any scheduled surgery that precludes compliance with treatment.
6. Known allergies to any of the ingredients of Papilocare®.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Study Population: Women over 18 years old with positive HPV with lesions in the cervical mucosa, and concordant colposcopy findings are eligible for the study.
Sampling Method: Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
The assessment of effectiveness of PAPILOCARE® in the regression of cervix cytological abnormalities caused by HPV. | Assessment at 6 months (or at 12 months)
  The percentage of patients with normalized cytology with respective colposcopy findings, as a change from ASCUS or LSIL to normal cytology supported by colposcopy.

SECONDARY OUTCOMES:
Assessment of ΗPV clearance | Assessment at 6 months (or at 12 months).
  The percentage of patients with complete or partial clearance of HPV confirmed by molecular HPV test (PCR or genetic diagnostic kits) that can detect High Risk (HR) strains.
The assessment of patient satisfaction level from treatment | Assessment at 6 months (or at 12 months).
  Changes in a 10-point satisfaction scale (0: "not satisfied at all", 10: "completely satisfied") from inclusion date.
The assessment of device safety | Treatment period (6 or 12 months).
  Recording of adverse events throughout the treatment period.

OTHER OUTCOMES:
The assessment of biopsy results (where available) | Assessment at 6 months (or at 12 months).
  The percentage of patients who improve and / or those who maintain the same degree of histological lesion at 6 months or 12 months from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Ginis, MD, Study Director — Elpen Pharmaceutical Co. Inc.
Locations (4):
- Greece (4):
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Larissa, Larissa
  - University General Hospital of Patra, Pátrai
  - "HIPPOKRATION" General Hospital of Thessaloniki, Thessaloniki

REFERENCES:
- [Background] Agorastos T, Chatzistamatiou K, Zafrakas M, Siamanta V, Katsamagkas T, Constantinidis TC, Lampropoulos AF; LYSISTRATA study group. Epidemiology of HPV infection and current status of cervical cancer prevention in Greece: final results of the LYSISTRATA cross-sectional study. Eur J Cancer Prev. 2014 Sep;23(5):425-31. doi: 10.1097/CEJ.0000000000000060. PMID 24977385
- [Background] Serrano L, Lopez AC, Gonzalez SP, Palacios S, Dexeus D, Centeno-Mediavilla C, Coronado P, de la Fuente J, Lopez JA, Vanrell C, Cortes J. Efficacy of a Coriolus versicolor-Based Vaginal Gel in Women With Human Papillomavirus-Dependent Cervical Lesions: The PALOMA Study. J Low Genit Tract Dis. 2021 Apr 1;25(2):130-136. doi: 10.1097/LGT.0000000000000596. PMID 33746195